CLINICAL TRIAL: NCT01490346
Title: A Compartmental Analysis of HIV Reservoirs and Immune Reconstitution
Brief Title: Tissue Drug Levels of HIV Medications
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0712M22448; P01AI074340 (NIH)
Record Dates: First submitted 2011-10-24; First posted 2011-12-13 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV 1; Pharmacokinetics; Drug levels; Treatment naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood & lymphatic tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ART treated individuals
  Interventions: Drug: Initiation of anti-retroviral therapy

INTERVENTIONS:
Drug: Initiation of anti-retroviral therapy — Subjects begin taking a preferred initial anti-retroviral regimens as determined by their primary care provider. Intracellular levels of those medications are measured.

SUMMARY:
The aim of this study is to find out why HIV continues to make copies in people taking HIV drugs. The investigators want to know if the medications most people use to treat HIV get into the lymphatic tissue where HIV persists.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Treatment naive or >30 days off ARV therapy
* Documented sensitivity to prescribed antiretrovirals
* Age ≥ 18 years
* Negative pregnancy test for eligible women of childbearing potential
* Ready to start ARV therapy

Exclusion Criteria:

* Contraindications to surgical & endoscopy procedures (as judged by PI)
* Psychiatric or psychological illness that would make adherence to protocol procedures unlikely
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive individuals beginning anti-retroviral treatment.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intracellular antiretroviral drug concentrations | Measured at baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months & 6 months

SECONDARY OUTCOMES:
Evidence of HIV replication in blood and lymphoid tissue | Measured at baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States